CLINICAL TRIAL: NCT06538480
Title: Open-Label Study of Zopapogene Imadenovec Retreatment and Vector Shedding Evaluation in Adult Patients With Recurrent Respiratory Papillomatosis
Brief Title: Zopa Retreatment and Vector Shedding in Adults With RRP
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Precigen, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRGN-2012-301
Record Dates: First submitted 2024-08-01; First posted 2024-08-05 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Recurrent Respiratory Papillomatosis; Papillomavirus Infection; Papillomaviridae
Keywords: Human Papilloma Virus; laryngotracheal disease; papillomatous disease; Viral Shedding; Retreatment; Zopapogene imadenovec
MeSH Terms: conditions — Recurrent respiratory papillomatosis; Papillomavirus Infections

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1 Vector Shedding (Experimental): Zopa administered subcutaneously at 5 × 10^11 particle units on Day 1, Week 2, Week 6, and Week 12. Samples for vector shedding to be collected from urine, feces, skin, and nasal tissue.
  Interventions: Drug: Zopapogene imadenovec (Zopa)
- Cohort 2 Retreatment (Experimental): Patients with prior treatment with Zopa (5 × 10^11 PU per injection) and require clinically indicated debulking procedure
  Interventions: Drug: Zopapogene imadenovec (Zopa)

INTERVENTIONS:
Drug: Zopapogene imadenovec (Zopa) — Zopa will be administered as 4 subcutaneous administrations over a 12-week interval.

SUMMARY:
This open-label study evaluates safety, vector shedding, and retreatment efficacy of Zopapogene imadenovec (Zopa) in adults with recurrent respiratory papillomatosis (RRP). Two cohorts will be enrolled (n=30): Cohort 1 to assess the magnitude and duration of adenoviral vector shedding in urine, feces, skin, and nasal tissue; Cohort 2 to assess the complete response rate following retreatment.

ELIGIBILITY:
Key Inclusion Criteria:

* Age 18 years and older.
* Clinical diagnosis of recurrent respiratory papillomatosis with histological confirmation of papilloma.
* Cohort 1: Treatment-naïve with respect to Zopa.
* Cohort 2: Received a minimum of four administrations of Zopa at 5 × 10^11 PU per injection and require clinically indicated debulking procedures.
* Presence of laryngotracheal papillomas accessible for endoscopic cleanout.
* ECOG performance status 0 or 1.
* Sexually active participants of reproductive potential must agree to use contraception during treatment and for 120 days for males and 6 months for females after last dose.
* Ability to understand and sign informed consent.

Key Exclusion Criteria:

* Conditions or therapies that increase risk or interfere with participation per investigator judgment.
* Systemic corticosteroids >10 mg prednisone equivalent or other immunosuppressive medications within 14 days prior to dosing.
* Other systemic RRP treatments or investigational agents within 30 days.
* History of heparin-induced thrombocytopenia or vaccine-induced thrombotic thrombocytopenia.
* Active uncontrolled HIV, hepatitis B, or hepatitis C infection.
* Pregnant or nursing women.
* Known allergy to any study drug component.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-07-11 (Actual); Primary Completion 2027-12-02 (Estimated); Study Completion 2028-12-02 (Estimated)

PRIMARY OUTCOMES:
Cohort 1 Vector shedding | Up to 6 weeks following last administration, with additional collections if needed until two consecutive measurements at or below limit of detection
  Magnitude and duration of Zopa vector shedding measured in urine, fecal, skin, and nasal tissue
Cohort 2 Complete Response Rate | 12 months following last administration
  Percentage of subjects achieving a complete response defined as no clinically indicated debulking procedures during the 12 months following completion of Zopa retreatment.

SECONDARY OUTCOMES:
Interval to First Debulking Procedure (Cohort 2) | 3 years following last administration
  Determine the interval to the first debulking procedure following retreatment with Zopapogene imadenovec (Zopa).
Safety and Tolerability of Zopa (Cohort 1 and Cohort 2) | Up to 28 days after last administration, with extended monitoring during follow-up.
  Assess the safety and tolerability of Zopa in adult subjects with recurrent respiratory papillomatosis (RRP), including incidence and severity of adverse events graded per CTCAE v5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Amy Lankford, PhD, Study Director — Precigen, Inc
Locations (3):
- United States (3):
  - Winship Cancer Institute, Emory University, Atlanta, Georgia
  - National Institute of Health, Bethesda, Maryland
  - University of Cincinnati, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: Undecided